CLINICAL TRIAL: NCT03506828
Title: The Effect of Adding Phenol With Fluoroscopy Guided Radiofrequency Ablation of T2-T3 Versus Thoracoscopic Sympathectomy in Palmar Hyperhidrosis.
Brief Title: Phenol With Fluoroscopy Guided Radiofrequency Ablation of T2-T3in Palmar Hyperhidrosis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MFM-IRB, MD/17.11.08
Record Dates: First submitted 2018-04-13; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Excessive Sweating of the Hands
MeSH Terms: interventions — Sympathectomy; Radiofrequency Ablation; Phenol

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single blind (Investigator) study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical sympathectomy (Active Comparator): All patients in this group will have standard surgical procedure
  Interventions: Procedure: Surgical sympathectomy
- Radiofrequency ablation with phenol injection (Active Comparator): patient will receive radiofrequency ablation of T2 and T3 sympathetic ganglia + phenol 6% (0.5ml) injection
  Interventions: Procedure: Radiofrequency ablation with phenol injection

INTERVENTIONS:
Procedure: Surgical sympathectomy — thoracoscopic sympathectomy
  Arms: Surgical sympathectomy
Procedure: Radiofrequency ablation with phenol injection — All patient in this group will have radiofrequency ablation of T2 and T3 sympathetic ganglia with phenol injection
  Arms: Radiofrequency ablation with phenol injection

SUMMARY:
Primary hyperhidrosis is a disorder characterized by excessive and chronic sweating in the absence of a sweating trigger. The disorder can be severe and interfere with normal daily activities of the patients.

The gold-standard treatment in severe cases of hyperhidrosis is thoracoscopic sympathectomy betweenT2 and T4. These procedures are regularly performed in surgical units under general anaesthesia which needs special anesthetic considerations which is complex and associated with a lot of complications.

Radiofrequency ablation of the sympathetic chain for treatment of hyperhidrosis is considered alternative to thoracoscopic sympathectomy. The procedure is safe, inexpensive and done under sedation with local anaesthesia in an outpatient setting, but its success rate is still significantly lower than endoscopic sympathectomy.

The purpose of this study is to determine whether adding phenol 6% in a mixture with glycerin will increase the efficacy of fluoroscopy guided radiofrequency ablation of T2, T3 sympathetic ganglia in hyperhidrosis in comparison to surgery without significant side effects to provide safe and effective method rather than surgery.

DETAILED DESCRIPTION:
Primary hyperhidrosis is a disorder characterized by excessive, chronic sweating in the absence of a sweating trigger. This condition must be differentiated from secondary hyperhidrosis, which is due to a lot of stimuli as infection, malignancy, drugs, anxiety, neurological and endocrine disorders.

Primary hyperhidrosis is caused by hyperactivity of the sympathetic system. The etiology of the disease is unknown and appears simultaneously. It affects patients between 15 and 40 years of age and may cause serious damage to their quality of life.

The first line of treatment of hyperhidrosis is non-surgical methods as topical antiperspirants, anti-cholinergic and Botox, but the disadvantages of this treatment are short term relieve, so repetition of this treatment is required.

Thoracoscopic Sympathectomy of the sympathetic chain between T2 and T4 is considered the gold-standard treatment in severe cases of hyperhidrosis. These procedures are performed in surgical units under general anaesthesia which needs special anesthetic considerations in the form of double lumen tube and one lung ventilation.

Complications like pneumothorax, surgical emphysema, lung injury, lobar collapse, atelectasis, pleural effusion; bleeding, Horner's syndrome and neuritis have been described. Postoperative pain is more severe which can occasionally require opiate analgesia.

Radiofrequency ablation of the sympathetic chain is considered alternative to thoracoscopic sympathectomy for hyperhidrosis. The procedure is safe, inexpensive and done under sedation with local anaesthesia in an outpatient setting, but its success rate is still significantly lower than endoscopic sympathectomy.

McCormack et al. concluded that there are anatomical variations in the position of sympathetic trunk which are thought to be one of the main causes of failure and patient dissatisfaction after thoracic sympathetic neurolysis in hyperhidrosis.

Previous studies tried to increase the efficacy of radiofrequency ablation of T2, T3 sympathetic ganglia in hyperhidrosis via adding alcohol 100% to cover the anatomical variations of the sympathetic trunk. Alcohol is intensely painful during injection, so large volume of local anaesthetics is injected prior to alcohol. Also, it is hypobaric, water soluble and spread rapidly from the injection site, so large volume is required. In addition, the incidence of neuritis is very high with its injection.

Phenol is primarily a local anesthetic at lower concentrations and becomes more neurolytic at higher concentration. Unlike alcohol, it is not painful on injection. It is prepared in a mixture with glycerin so it is highly soluble and hyperbaric and diffuses slowly into the local tissues.

In this study, the effect of adding phenol 6% with percutaneous fluoroscopy guided radiofrequency ablation of T2, T3 sympathetic ganglia in hyperhidrosis will be evaluated. The study hypothesizes that adding phenol 6% in a mixture with glycerin will increase the efficacy of radiofrequency ablation of T2, T3 sympathetic ganglia in hyperhidrosis in comparison to surgery without significant side effects to provide safe and effective method rather than surgery for hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status grades I and II

Exclusion Criteria:

* Patient refusal.
* Hepatic impairement.
* Renal impairment.
* Neuromuscular diseases.
* History of opioid abuse.
* Coagulopathies.
* Cardiovascular diseases.
* Respiratory diseases.
* Previously failed cases either after percutaneous or thoracoscopic sympathectomy.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2020-01-02 (Estimated)

PRIMARY OUTCOMES:
Temperature of the ipsilateral palm of the hand | For six months after the procedure

SECONDARY OUTCOMES:
Postoperative pain scores | For 24 hours after the procedure
  The level of pain based on visual analog scale (VAS) (where 0= no pain and 10= worst pain) will be assessed
postoperative cumulative analgesic consumption | For 24 hours after the procedure
  Total amount of post-operative analgesics (ketorolac and fentanyl) will be recorded.
Occurrence of pneumothorax | immediately after the procedure
  Patients will be transferred to the PACU and chest x ray will be done to exclude pneumothorax.
Severity of compensatory hyperhidrosis | For six months after the procedure
  Compensatory hyperhidrosis defined as excessive sweating after the procedures in areas of the body that previously did not sweat mainly in axilla, back, and lower limbs and will be assessed and classified into 4 degrees Not present, Mild Sometimes noticeably sweaty and sometimes not sweaty, Moderate Always aware but not troublesome, or troublesome but controlled by clothing, and Sever Causes embarrassment
Patient satisfaction | For six months after the procedure
  Patient satisfaction with their procedure will be measured with a four-grade scale: 0 (not satisfied), 1 (slightly satisfied), 2 (satisfied) and 3 (very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Gamal M El Morsy, MD, Study Chair — Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided